CLINICAL TRIAL: NCT06974630
Title: Cervical Erector Spinae Plane Block vs Cervical Plexus Block in Controlling Acute Postoperative Pain After Thyroidectomy: A Randomized Controlled Study
Brief Title: Cervical Erector Spinae Plane Block vs Cervical Plexus Block in Controlling Acute Postoperative Pain After Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Elsaid Abdel Fattah, Lecturer of Anesthesia, Surgical ICU and Pain Management, Faculty of Medicine, National Cancer Institute, Cairo University, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP2411-501-102-193
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Cervical; Erector Spinae Plane Block; Cervical Plexus Block; Postoperative Pain; Thyroidectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Cervical Plexus Block

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB group (Experimental): Patients will receive bilateral ultrasound-guided cervical erector spinae plane block using 15 ml of bupivacaine 0.25% on each side.
  Interventions: Other: Cervical erector spinae plane block
- SCPB group (Active Comparator): Patients will receive bilateral ultrasound-guided superficial cervical block using 15 mL of 0.25% plain bupivacaine on each side of the neck.
  Interventions: Other: Cervical plexus block

INTERVENTIONS:
Other: Cervical erector spinae plane block — Patients will receive bilateral ultrasound-guided cervical erector spinae plane block using 15 ml of bupivacaine 0.25% on each side.
  Other Names: Bupivacaine 0.25%
  Arms: ESPB group
Other: Cervical plexus block — Patients will receive bilateral ultrasound-guided superficial cervical block using 15 mL of 0.25% plain bupivacaine on each side of the neck.
  Other Names: Bupivacaine 0.25%
  Arms: SCPB group

SUMMARY:
This study aims to compare the efficacy and safety of cervical erector spinae plane block vs. cervical plexus block in controlling acute postoperative pain after thyroidectomy.

DETAILED DESCRIPTION:
Thyroidectomy is one of the most commonly performed surgeries in females worldwide, as thyroid disease predominantly affects females with a ratio of 4:1. Thyroid operations can cause mild to moderate incisional pain. It has also been reported that the morphine consumption on the first postoperative day is 90%.

Cervical plexus block, either superficial or deep or combinations given bilaterally, could easily lead to an adequate block appropriate for thyroid surgery without any significant side effects.

Erector spinae plane block (ESPB) is the new favorite among various fascial plane blocks. Local anesthetic drug is injected in the fascial plane superficial to the transverse process and deeper to the erector spinae muscle (ESM).

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both genders.
* American Society of Anesthesiologists (ASA) physical status I-II.
* Scheduled for either hemi- or total thyroidectomy.

Exclusion Criteria:

* Known allergy to local anesthetics.
* Allergy to all opioid medications.
* Pregnant patient.
* Previous neck surgery.
* Recent use of non-steroidal anti-inflammatory drugs (NSAIDs), opioids or steroid injection within 2 weeks.
* Those who cannot utilize the numeric rating scale (NRS) .
* Chronic opioid use.
* Coagulopathy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 48 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the numeric rating scale (NRS) > 3 to be repeated after 30 min if pain persists until the NRS < 4.

SECONDARY OUTCOMES:
Time to the 1st rescue analgesia | 48 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to first dose of morphine administrated).
Intraoperative fentanyl consumption | Intraoperatively
  Additional bolus doses of fentanyl 1 µg/kg will be given if the mean arterial blood pressure (MAP) or heart rate (HR) rises above 20% of baseline levels.
Degree of pain | 48 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at post-anesthesia care unit (PACU), 1, 2, 4, 6, 8, 12, 18, 24, 36 and 48 h postoperative.
Incidence of adverse events | 48 hours postoperatively
  Incidence of adverse events such as nausea, vomiting, hypotension, bradycardia, cough, bronchospasm, and sore throat will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.